CLINICAL TRIAL: NCT02007967
Title: Can Non-Contrast Magnetic Resonance Angiography Accurately Define Arterial Access and Aortic Root Anatomy in Patients Referred for Transcatheter Aortic Valve Implantation?
Brief Title: Non-Contrast Magnetic Resonance Angiography Assessment of Patients Referred for Transcatheter Aortic Valve Implantation
Status: Terminated | Type: Observational
Why Stopped: Difficulty enrolling patients
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Troy LaBounty, Assistant Professor, Internal Medicine, University of Michigan
Other Study IDs: HUM00070087
Record Dates: First submitted 2013-11-08; First posted 2013-12-11 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of this proposal is to examine the feasibility and accuracy of non-contrast magnetic resonance angiography (MRA) to comprehensively evaluate individuals referred for transcatheter aortic valve implantation (TAVI).

ELIGIBILITY:
Inclusion Criteria:

* Adults with severe aortic stenosis referred for possible transcatheter aortic valve implantation with clinically indicated computed tomography imaging

Exclusion Criteria:

* Inability or unwillingness to consent
* Inability to complete magnetic resonance imaging (MRI) study
* Contraindication to MRI
* Participation in another research study
* Non-diagnostic computed tomography scan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will include patients undergoing clinically indicated computed tomography angiography for evaluation for possible transcatheter aortic valve implantation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Minimal luminal size for aorta and ileofemoral arteries | 3 hours
  Compare luminal diameter for each segment of the ileofemoral arteries and aorta between MRI and CT

SECONDARY OUTCOMES:
Graded image quality | 3 hours
  Compare graded image quality for ileofemoral arteries, aorta, and aortic annulus between MRI and CT
Annular size | 3 hours
  Compare annular diameter, area, and perimeter between MRI and CT

CONTACTS AND LOCATIONS:
Overall Officials: Troy M LaBounty, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cardiovascular Center, Ann Arbor, Michigan, United States